CLINICAL TRIAL: NCT07325578
Title: Evaluation of the Epione Robotic System for Image-guided Percutaneous MSK Procedures of the Pelvis and Spine in USA. A Prospective Study on Feasibility, Safety and Accuracy
Brief Title: U.S. Prospective Evaluation of EPIONE Device for Percutaneous MSK Procedures
Acronym: EPIOS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Quantum Surgical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CA-BO-CIP-0130
Record Dates: First submitted 2025-12-19; First posted 2026-01-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Bone Tumor; Osteoporosis; Traumatic Fracture
Keywords: percutaneous procedure; robot assistance; bone procedure
MeSH Terms: conditions — Bone Neoplasms; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- CT guidance (Experimental): The procedure is performed under CT guidance.
  Interventions: Device: Percutaneous procedure in the MSK structures of the pelvis and/or the spine
- CBCT guidance (Experimental): The procedure is performed under CBCT guidance.
  Interventions: Device: Percutaneous procedure in the MSK structures of the pelvis and/or the spine

INTERVENTIONS:
Device: Percutaneous procedure in the MSK structures of the pelvis and/or the spine — The introducer placement is performed with the Epione device.

SUMMARY:
The goal of this investigational device exemption is to evaluate the Epione assistance for introducer placement during percutaneous procedures in musculo-skeletic (MSK) structures of the pelvis and the spine in adults.

The main question is the determination of the rate of feasible procedures assisted by the Epione device

Participants will undergo their procedure(s) as planned by their physician. If they accept to participate to the study, the differences with standard of care will be:

* The use of the Epione device to place the introducer(s), instead of freehand placement if they do not participate
* Additional CT or CBCT scans during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥22 years old,
* Patients approved for CT- or CBCT-guided MSK procedure in the pelvis or spine (except the cervical area) under general anesthesia,
* Patients who have signed an IRB-approved informed consent form
* Patients approved for coverage by their insurance for routine costs involved in this standard of care procedure
* Inclusion criteria linked to the freehand procedure have been discussed and validated

Exclusion Criteria:

* Patients with contraindication to undergo general anesthesia,
* Patients unable to maintain appropriate breathing control,
* Patients requiring CT- or CBCT-guided percutaneous procedure on target areas other than those indicated
* Patients unable to fully understand all relevant aspects of the clinical study necessary for their decision to participate, or who could be manipulated or unduly influenced because of a compromised position, expectation of benefits or fear of retaliatory response,
* Pregnant or breast-feeding women,
* Patients subject to a legal protection measure,
* Patients already participating in another conflicting interventional clinical study,
* Patients for whom the scan field of view cannot contain the anatomy of interest, the overlaying skin surface, skin markers and the whole patient reference.
* Patients having a coagulation abnormalities or bleeding disorder
* Patients having an active infection on the day of intervention
* Patients having a history of previous surgery resulting in an existing hardware precluding percutaneous approach
* Exclusion criteria linked to the freehand procedure have been discussed and validated

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Feasability | 5 months
  Rate of successful insertions of the introducer with the assistance of the Epione device.

SECONDARY OUTCOMES:
Safety Adverse Event | 6 months
  Adverse event(s) (AE): all AEs (serious and non-serious, related and not related to the device or the procedure(s))
Accuracy | 5 months
  Lateral and 3D deviations, being the distance (mm) between the tip of the inserted introducer in its final position and its orthogonal projection on the first planned trajectory (lateral deviation) and the distance (mm) between the tip of the inserted introducer in its final position and the tip of the first planned trajectory (3D deviation).

CONTACTS AND LOCATIONS:
Overall Officials: Sean Tutton, MD, Principal Investigator — UC San Diego
Locations (3):
- United States (3):
  - UC San Diego, San Diego, California
  - Baptist Hospital Of Miami, Inc, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Age, Sex, Ethnicity, Race will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: by the end of the study
Access Criteria: everyone, they will be described in the report and publication